CLINICAL TRIAL: NCT06919744
Title: Direct Intracranial Venous Stenting Evaluation in Patients With Idiopathic INtracranial Hypertension in the Early Phase
Brief Title: Intracranial Venous Stenting Evaluation in Patients With Idiopathic Intracranial Hypertension in the Early Phase
Acronym: DIVE IIN EARLY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Ministère de la Santé (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL 23_0430; 2024-A02444-43 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Intracranial Hypertension (IIH)
Keywords: Intracranial hypertension; papillary edema; stenting; transverse sinus vein; chronic headache; tinnitus
MeSH Terms: conditions — Pseudotumor Cerebri; Intracranial Hypertension; Headache Disorders; Tinnitus | interventions — Acetazolamide; Methods; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- best medical care (Active Comparator): Acetazolamide and recommended weight loss
  Interventions: Drug: Best medical care
- Experimental (stenting, neuro-radiological intervention) (Experimental): Stenting of the tranverse sinus vein
  Interventions: Device: Intervention (stenting)

INTERVENTIONS:
Drug: Best medical care — Acetazolamide will be introduced at the time of papilledema discovery. Weight loss will be recommended.
  Other Names: Acetazolamide; Weight loss
  Arms: best medical care
Device: Intervention (stenting) — Transverse venous sinus will be stented by neuro-radiological intervention
  Arms: Experimental (stenting, neuro-radiological intervention)

SUMMARY:
This study is aimed at patients suffering from recently discovered intracranial hypertension, caracterized by visual loss, chronic headache and/or tinnitus. The goal is to evaluate if stenting of a specific vein in the brain could decrease the hypertension and improve associated symptoms. Patients will be randomly assigned in either best medical care group (recommended medication associated with weight loss) or interventional group (best medical car + stenting of the specific vein) and will undergo specific follow-up visits after 1, 3 and 12 months.

DETAILED DESCRIPTION:
The DIVE-IIN-EARLY trial is a multicenter randomized controlled trial designed to evaluate whether transverse venous sinus stenting is more effective than best medical therapy alone as first-line treatment for patients with idiopathic intracranial hypertension (IIH). The study targets patients with a new diagnosis of IIH with bilateral transverse sinus stenosis or unilateral stenosis of the dominant transverse sinus with a hypoplastic contralateral sinus.

Idiopathic intracranial hypertension is, in most cases, associated with narrowing of the transverse sinus vein, which may be the cause of increased intracranial blood pressure, resulting in the accumulation and increase in intracranial fluid pressure. This increased pressure is thought to be responsible for papilledema, chronic headaches, and tinnitus, among other symptoms.

Restoring a normal luminal diameter of the transverse sinus using a stent could therefore allow for the rapid restoration of normal intracranial pressures and an improvement in various symptoms.

Stent implantation in the transverse sinus is now part of standard care, but no large-scale clinical trial has formally established the superiority of the technique compared to the standard of care (drug therapy combined with weight gain). This study aims to provide evidence on the potential benefits of transverse venous sinus stenting as a treatment option for patients with idiopathic intracranial hypertension, which could significantly change the current management approach to this disease.

Usual medication for this condition is acetazolamide, but it's efficacy as well as it's tolerance is mostly poor. By proposing stenting in the early phase of the disease, one could avoid long term symptoms such as loss of vision and chronic headache.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old at inclusion.
2. Subject with definite new diagnosis (˂ 3 months) of IIH satisfying the modified Dandy criteria (A to E)
3. Subject with intracranial TVS stenosis on dominant transverse sinus and hypoplastic contralateral one (or bilateral TVS stenosis) diagnosed on MRI
4. Normal MRI findings excepted intracranial TVS stenosis or IIH related abnormalities
5. Subject with ophthalmologic IIH symptoms and signs (RNFL ≥ 130 µm, Frisen score ≥ 2, and absence of differential diagnostic)
6. Subject without macular ganglion cells atrophy seen on OCT
7. Patient having received information about data collection and having signed and dated an Informed Consent Form
8. Subjects must be able to attend all scheduled visits and to comply with all trial procedures
9. Subjects must be covered by public health insurance

Exclusion Criteria:

1. Subject previously treated with acetazolamide for IIH
2. Known contrast product, Nickel, titanium allergy
3. Exposure to an oral drug, substance, or disorder that has been associated with elevation of intracranial pressure within 2 months of diagnosis (lithium, vitamin A, tetracycline and related compounds)
4. History of intracranial venous thrombosis or intracranial neoplasia
5. Fulminant decrease of visual acuity due to the IIH defined as a visual loss (of the most seriously impaired eye) of at least 3/10 (from corrected vision) within 4 weeks, in absence of any other ophthalmologic pathology and Mean Deficit of visual field superior to -10 dB
6. Macular ganglion cells atrophy seen on OCT
7. Optic nerve atrophy
8. Amblyopia
9. Refractive error greater ±8 sphere or more than ±3 in cylinder in either eye if there are abnormalities in funduscopy (optic disc tilt, staphyloma), previous glaucoma, other disorders causing visual loss
10. Pregnancy: if a woman is of childbearing potential a urine or serum beta HCG test is positive
11. Patient with a severe or fatal comorbidity that will likely prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.
12. Evidence of intracranial hemorrhage (subarachnoid hemorrhage (SAH), intracerebral hemorrhage (ICH), etc.)
13. Life expectancy under 6 months
14. Chronic IIH
15. Patients with renal failure (creatinine > 1.5 mg/dl and/or creatinine clearance < 60 mL/min, except if patient is already on hemodialysis)
16. History of previously implanted intra-cranial sinus stent
17. Previous gastric bypass surgery
18. Contra-indication to general anesthesia
19. Contra-indication to aspirin, clopidogrel or other P2Y12 anti-aggregant
20. History of chronic obstructive pulmonary disease or other severe respiratory disease
21. History of deep vein thrombosis or pulmonary embolism
22. History of atrial fibrillation or other risks of stroke
23. Cerebral vascular lesions (arteriovenous malformation, arteriovenous fistula, aneurysms, significant stenosis of extra- or intra-cranial vessels other than the targeted venous sinus stenosis, intracranial artery dissection, etc.).
24. Anatomical anomaly of the venous sinus which would prevent safe catheterization and stenting
25. Subject who are in a dependency or employment with the sponsor or the investigator
26. Participation in another clinical trial or administration of an unapproved drug within the last 4 weeks before the screening date
27. Subject protected according to the French Public Health Code (e.g. patients under law protection, prisoners, pregnant, parturient or lactating women, and patients under guardianship/curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with resolved papilledema and normalization of intra-cranial pressure | 3 months
  Rate of patients with resolved papilledema (defined as Frisén scale grade 0-1 on OCT, without ganglion cells damage, and RNFL ˂ 130 µm) and normalization of intra-cranial pressure (defined as ≤ 25 cm H20 or 18 mmHg measured on lumbar puncture) at 3 months. Papilledema will be studied in the most affected eye.

SECONDARY OUTCOMES:
HIT-6 grading scale score | 3 and 12 months
  Change in mean HIT-6 grading scale score (patient's questionnaire containing 6 questions to evaluate the severity of headache)
Monthly headache days | 3 and 12 months
  Change in monthly headache days (within the last month) reported on patients' dairy
THI score | 3 and 12 months
  Change in THI (Tinnitus Handicap Inventory) score
Visual field | 3 and 12 months
  Change in decibel of Mean Deficit visual field assessed on automated perimetry in both eyes with Humphrey Field Analyzer SITA Standard 24-2 test pattern. Each participant will have at least 2 initial visual field examinations conducted at least 30 minutes apart. The 2 Perimetric Mean Deviation (PMD) measurements will be averaged.
Visual acuity | 3 and 12 months
  Change of visual acuity score evaluated on ETDRS (far vision) at 4 meters and reproducible lighting, and Parinaud scale (near vision) using the best optical correction
Papilledema | 3 and 12 months
  Change of papilledema assessed on Frisen score and RNFL on OCT
Patient's autonomy | 3 and 12 months
  Change in quality of life assessed on EQ5D questionnaire
Patient's cognition | 12 months
  Change in Montreal Cognitive Assessment (MoCA)
Cognition | 12 months
  Change in Trail Making Test (TMT) A and B

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Montpellier Hôpital Gui de Chauliac, Montpellier
  - CHU de REIMS, Reims
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No